CLINICAL TRIAL: NCT03751735
Title: Evaluation of the Efficacy for Two Doses of Intracavernous Injection of Wharton Jelly Stem Cells for the Treatment of Diabetic Erectile Dysfunction
Brief Title: Efficacy of Wharton Jelly in Erectile Dysfunction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sophia Al-Adwan (Other)
Responsible Party: Sponsor-Investigator, Sophia Al-Adwan, Researcher, Clinical coordinator, University of Jordan
Organization: University of Jordan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WJEF.EDUJCTC
Record Dates: First submitted 2018-11-13; First posted 2018-11-23 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Erectile Dysfunction Associated With Type 2 Diabetes Mellitus
Keywords: Diabetes; Wharton jelly mesenchymal stem cells; efficacy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose 1 (Experimental): Dose I of Wharton Jelly Mesenchymal stem cells (WJ-MSC) Two intracavernous injections of 20 million of WJ-MSC cells will be given to erectile dysfunction patients at baseline and 4th week of follow up
  Interventions: Biological: Wharton Jelly Mesenchymal stem cells

INTERVENTIONS:
Biological: Wharton Jelly Mesenchymal stem cells — Intracavernous injection of Wharton Jelly Mesenchymal stem cells.

SUMMARY:
Efficacy of Intracavernous injection of Wharton jelly Mesenchymal stem cells for the treatment of erectile dysfunction in diabetic patients.

DETAILED DESCRIPTION:
This study will be conducted at the Cell Therapy Center (CTC), Jordan, in which 22 male patients ranging from 25-70 years diagnosed with erectile dysfunction will be selected. This diagnosis is based on medical history, validated questionnaires, physical examinations, laboratory tests and specific diagnostic tests.

The patients are followed by clinical assessment, laboratory investigations as well as Doppler ultrasound.

The investigators hypothesize that the intracavernous injection of stem cells will facilitate the recovery of erectile function resulting in satisfying clinical outcomes in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male patients ranging from 25 to 70 years.
2. History of chronic erectile dysfunction for at least six months.
3. Baseline international index of erectile function (IIEF) score of < 26.
4. Not interested or able to use phosphodiesterase type 5 inhibitor (PD5i) drug therapy and willing to forgo theses treatments for the first 6 month period following study treatment.
5. Body Mass Index between 20-30.
6. Willing to provide written informed consent, complete questionnaire, and to be available for all baseline treatment and follow up examinations required by protocol.

Exclusion Criteria:

1. Current urinary tract or bladder infection.
2. Clinical/Laboratory evidence of transmissible diseases.
3. Clinically evident penile anatomical deformities(e.g., Peyronie's disease) or history of priapism.
4. Skin irritation, infection, wound, sore or disruption in the immediate areas of skin entry for penile injection.
5. Current or previous malignancy.
6. Use of any non study treatment for erectile function within 4 weeks of study treatment.
7. Lack of willingness to continue through 6 months after study treatment.
8. Any previous penile implant or penile vascular surgery.
9. Uncontrolled hypertension or hypotension(systolic blood pressure > 170 or < 90 mm Hg, and diastolic blood pressure > 100 or < 50 mm Hg).
10. Reported unstable cardiovascular disease (e.g., unstable angina, myocardial infarction within past 6 months, cardiac failure or life-threatening arrhythmia, congestive heart failure) or symptomatic postural hypotension within 6 months before screening.
11. Bleeding or clotting disorder, use of anticoagulant therapy.
12. Lab values for complete blood count (CBC), prothrombin time (PT)/ partial thromboplastin time (PTT)/ international normalized ratio (INR), alanine aminotransferase (ALT), aspartate aminotransferase (AST) and creatinine falling outside the normal lab values.
13. Systemic autoimmune disorder.
14. Significant active systemic or localized infection.
15. Receiving immunosuppressant medications.
16. Post-radical prostatectomy.

Ages: 25 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2019-01-13 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Assessment of the efficacy of injecting Wharton Jelly derived Mesenchymal Stem Cells by Penile Doppler ultrasonography. | 12 months
  Patients will be evaluated for the efficacy of the intracavernous injection of Wharton Jelly derived Mesenchymal Stem Cells by Penile Doppler ultrasonography in which peak systolic velocity of the cavernosal arteries will be measured.
Assessment of the efficacy of injecting Wharton Jelly derived Mesenchymal Stem Cells by SHIM/IIEF/EHS questionnaires | 12 months
  The efficacy of the intracavernous injection of Wharton Jelly will be evaluated by scoring the SHIM/IIEF/EHS questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Abdalla Awidi, MD, Study Director — Cell Therapy Center
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided